CLINICAL TRIAL: NCT01961752
Title: The Efficacy of Topical Bupivacaine and Triamcinolone Acetonide Injection in the Relief of Pain After Endoscopic Submucosal Dissection for Gastric Neoplasia: A Randomized Double-blind, Placebo-controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2012-0147
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Gastric Cancer; Gastric Adenoma
Keywords: bupivacaine,; triamcinolone acetonide,; endoscopic; submucosal; dissection; Patients
MeSH Terms: conditions — Stomach Neoplasms | interventions — Sodium Chloride; Bupivacaine; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (Placebo Comparator)
  Interventions: Drug: Saline
- Bupivacaine only group (Experimental)
  Interventions: Drug: Bupivacaine + saline
- Bupivacaine with triamcinolone group (Active Comparator)
  Interventions: Drug: Bupivacaine + triamcinolone acetonide

INTERVENTIONS:
Drug: Saline — All patients undergo endoscopic submucosal dissection. The local injection was performed using 15 ml saline just before the ESD was finished. It was delivered through the endoscopy suite and injected into the cautery ulcer base in aliquots of 1 mL at equal intervals (1 cm apart). The number of injections per patient was dependent on the size of resection.
  Arms: Control group
Drug: Bupivacaine + saline — All patients undergo endoscopic submucosal dissection. The local injection was performed using a mixture of 10 ml bupivacaine (total 50 mg) and 5 ml saline just before the ESD was finished. It was delivered through the endoscopy suite and injected into the cautery ulcer base in aliquots of 1 mL at equal intervals (1 cm apart). The number of injections per patient was dependent on the size of resection.
  Arms: Bupivacaine only group
Drug: Bupivacaine + triamcinolone acetonide — All patients undergo endoscopic submucosal dissection. The local injection was performed using a mixture of 10ml bupivacaine (total 50 mg) and 5 ml triamcinolone acetonide (total 50 mg) just before the ESD was finished. It was delivered through the endoscopy suite and injected into the cautery ulcer base in aliquots of 1 mL at equal intervals (1 cm apart). The number of injections per patient was dependent on the size of resection.
  Arms: Bupivacaine with triamcinolone group

SUMMARY:
Although pain is a common complication of endoscopic submucosal dissection (ESD), management strategies are inadequate. bupivacaine is used for visceral pain control in chronic pain and in pain associated with surgery in clinical practice. Further, triamcinolone, a type of steroid, is often mixed with bupivacaine to lengthen the analgesic effect. The aim of this study was to evaluate the efficacy of topical bupivacaine and triamcinolone acetonide for abdominal pain relief and as a potential method of pain control after ESD for gastric neoplasia. We hypothesized that topical bupivacaine and/or triamcinolone acetonide injection after ESD would be effective for pain relief. For this, we designed randomized, double-blind, placebo-controlled trial. Eligible patients with early gastric neoplasm were randomized into one of three groups: bupivacaine (BV) only, bupivacaine with triamcinolone (BV-TA), or placebo. To evaluate the pain after ESD, the Present Pain Intensity (PPI) score and the Short-Form McGill Pain Questionnaire (SF-MPQ) were used to evaluate pain at 0, 6, 12 and 24 h after ESD.

ELIGIBILITY:
Inclusion Criteria:

* Age, between 20 and 80
* Patients who were scheduled to undergo ESD for gastric epithelial neoplasm at Severance Hospital between July 2012 and April 2013

Exclusion Criteria:

* Not providing written informed consent
* A history of any cardiac arrhythmias
* Current or regular use of analgesic medication for other indications
* Known other disease such as peptic ulcer disease or reflux esophagitis which could induce upper gastrointestinal pain
* Multiple lesions requiring ESD in a single patient
* Evidence of infectious disease or antibiotics therapy within 7 days prior to enrollment
* Participation in another clinical trial within 30 days prior enrollment
* Current pregnancy or breast feeding.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Present Pain Intensity (PPI) score | at 6 hour after endoscopic submucosal dissection (ESD)
  Present Pain Intensity (PPI) score at 6 hour after endoscopic submucosal dissection (ESD) is assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Severnace Hospital, Yonsei University Health System, Seoul, South Korea

REFERENCES:
- [Background] Kiriyama S, Oda I, Nishimoto F, Mashimo Y, Ikehara H, Gotoda T. Pilot study to assess the safety of local lidocaine injections during endoscopic submucosal dissection for early gastric cancer. Gastric Cancer. 2009;12(3):142-7. doi: 10.1007/s10120-009-0514-y. Epub 2009 Nov 5. PMID 19890693
- [Derived] Kim B, Lee H, Chung H, Park JC, Shin SK, Lee SK, Lee YC. The efficacy of topical bupivacaine and triamcinolone acetonide injection in the relief of pain after endoscopic submucosal dissection for gastric neoplasia: a randomized double-blind, placebo-controlled trial. Surg Endosc. 2015 Mar;29(3):714-22. doi: 10.1007/s00464-014-3730-4. Epub 2014 Jul 25. PMID 25060683